CLINICAL TRIAL: NCT06062004
Title: Evaluation of Different Lenticule Diameters in Myopic Astigmatism Correction With SMILE Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al Watany Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REF-2018-003
Record Dates: First submitted 2023-07-12; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Refractive Errors; Myopic Astigmatism
Keywords: SMILE; Myopia; Refractive Surgery; Astigmatism; Small Incision Lenticule Extraction
MeSH Terms: conditions — Refractive Errors; Astigmatism; Myopia

STUDY DESIGN:
Intervention Model Description: Hospital-based, comparative, prospective, interventional contralateral eye study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): group A, SMILE procedure with lenticule diameter of 6.5 mm
  Interventions: Procedure: Small Incision Lenticule Extraction (SMILE)
- Study cases (Active Comparator): group B, SMILE procedure with lenticule diameter of 7.0 mm
  Interventions: Procedure: Small Incision Lenticule Extraction (SMILE)

INTERVENTIONS:
Procedure: Small Incision Lenticule Extraction (SMILE) — All surgeries will be performed under topical anesthesia using the VisuMax femtosecond laser with the following parameters:
  * Cap thickness of 120 μm
  * Cap diameter of 1 mm larger than the lenticule diameter
  * Cap side cut angle 70°
  * 3 mm incision positioned at 100° and angled at 45°
  * Transition zone of 0.1 mm and clearance of 0.5 mm
  * Lenticule side cut angle of 90° and edge lenticule thickness of 15 μm

SUMMARY:
Small incision lenticule extraction (SMILE) is a refractive intrastromal procedure for myopia and myopic astigmatism correction. Most of the studies evaluating astigmatic correction by SMILE reported astigmatic under-correction, especially in high degrees of astigmatism.

This under-correction could be due to: first, the active eye tracker or the iris registration is not yet available to overcome the cyclotorsion that occurred during the treatment with the VisuMax femtosecond laser system (Carl Zeiss Meditec, Jena, Germany) which could be overcome by manual compensation technique, especially in higher degrees of cylinders (> 1.5 diopters (D)). Second, in patients with small lenticule diameters, the more abrupt change in thickness at the edge of the treated area could induce more stromal and epithelial healing in this area. Thus, the astigmatic correction would be less effective with small than large lenticule diameters for similar high preoperative astigmatism.

This study assessed the outcome of using a 0.5 millimeter (mm) larger lenticule diameter in the fellow eyes of myopic astigmatic correction SMILE participants. This assessment included the safety and effectiveness indices, the refractive and visual outcomes, the contrast sensitivity, and some morphological outcomes such as corneal curvature and epithelial and corneal thickness.

DETAILED DESCRIPTION:
Study Title: Evaluation of different lenticule diameters in myopic astigmatic correction with SMILE procedures Primary Investigator: Dr. Ahmed Sedky (Eye Subspecialty Center, Cairo, Egypt, 18 Elkhalifa Elmamoun Street, Heliopolis, Cairo, Egypt) Co-Investigators: Sherine S Wahba, Maged M Roshdy, Nermeen A Refaat Study Objectives Primary Objective: To study the effect of changing the lenticule diameter on the safety and effectiveness of myopic astigmatism correction with the SMILE procedure.

Secondary Objective: To compare other outcomes such as visual outcomes including immediate visual acuity, contrast sensitivity, and epithelial remodeling.

Participants and Methods:

Study Setting: Eye Subspecialty Center, Cairo, Egypt, 18 Elkhalifa Elmamoun Street, Heliopolis, Cairo, Egypt and Al Watany Eye Hospital, Althawra Street, Cairo, Egypt Study design: Hospital-based, comparative, prospective, interventional contralateral eye study Sample size and randomization: 50 participants fulfilling the inclusion criteria will be enrolled in the study. Their right eyes undergo SMILE procedure using the standard 6.5 mm lenticule diameter and their left eyes undergo SMILE procedure but using a larger lenticule diameter of 7.0 mm.

Ethical issues:

Institutional ethics committee approval will be obtained. Participants' informed consent will be taken and the procedure explained to them in their own language. Any intra-operative or post-operative complications occurring in either group will be documented and duly informed to the ethics committee

Preoperative evaluation:

1. Anterior and posterior segment clinical examination
2. Uncorrected distance visual acuity (UDVA) in decimal and logMAR units
3. Corrected distance visual acuity (CDVA) in decimal and logMAR units
4. Corneal tomography using the Pentacam high resolution (HR) (Oculus Optikgeräte, Wetzlar, Germany) including the flattest and steepest meridians (in keratometric diopters (D), the axes (in degrees)
5. Contrast sensitivity (CSV1000E test (Good-Lite, Elgin, Illinois, USA)) in 4 different special frequencies
6. Anterior segment Optical Coherence Tomography (Cirrus, Carl Zeiss Meditec, Jena, Germany) measurement of total corneal and epithelial thickness in µm Study duration: 3 months for recruitment of the patients.

Surgical technique:

All surgeries will be performed under topical anesthesia using the VisuMax femtosecond laser with the following parameters:

Cap thickness of 120 μm Cap diameter is either 7.5 mm for lenticule diameter 6.5 mm or 8.0 mm for lenticule diameter 7.0 mm.

Cap side cut angle 70° 3 mm incision positioned at 100° and angled at 45° A transition zone of 0.1 mm and clearance of 0.5 mm Lenticule side cut angle of 90° and edge lenticule thickness of 15 μm Directly preoperative, the limbus will be marked in the 0° to 180° axis with a marker pen in the upright head position on the slit lamp. Then, the patient will be positioned under the VisuMax femtosecond laser and instructed to look into the green flashing fixation light. Once proper centration is achieved, the eye will be docked to the patient interface and suction will be applied.

Manual compensation will be done by gently rotating the contact glass to align the horizontal marks on the eye to the 0° to 180° axis. Once both are aligned, the laser process will be done to create the refractive lenticule followed by its dissection and washing of the interface by a balanced salt solution.

Medication: will be the standard treatment; topical steroids and antibiotics 4 times per day for 10 days and tear substitutes 4 times daily for one to two months.

Postoperative evaluation:

Follow-up of the subjects will be done in 1 day, 1 week, 3 months, and 6 months.

Data will be collected for analysis starting from 1 week, including:

1. Uncorrected distance visual acuity (UDVA) in decimal and logMAR units
2. Corrected distance visual acuity (CDVA) in decimal and logMAR units
3. Corneal tomography using the Pentacam HR (Oculus Optikgeräte GmbH, Wetzlar, Germany) including the flattest and steepest meridians (in diopters (D), the axes (in degree)
4. Contrast sensitivity (CSV1000E test (Good-Lite, Elgin, IL, USA)) in 4 different special frequencies
5. Anterior segment Optical Coherence Tomography (Cirrus HD-OCT, Carl Zeiss Meditec, Jena, Germany) measurement of total corneal and epithelial thickness in µm.

ELIGIBILITY:
Inclusion Criteria:

* Age groups between 18 and 50 years
* Myopic astigmatism with up to -10.00 D spherical equivalent (SE) and a minimum astigmatism of -1.0 D and a maximum of -5 D. The astigmatism will be divided into low astigmatism (<0.75 D), moderate astigmatism (1.5- 3 D) and high astigmatism (>3 D).
* Corrected distance visual acuity (CDVA) of 0.7 or better (decimal)

Exclusion Criteria:

* Thin corneas (< 490 μm)
* Proven or suspicious cases of corneal ectatic conditions by corneal tomography
* Previous ocular surgeries
* Patients taking systemic steroids, immunosuppressants, oral contraceptives, or antidepressants
* Pregnant females
* Corneal scars or any ocular pathology likely to affect visual outcomes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
The safety index of using 7 and 6.5 mm lenticule diameters SMILE to treat myopic astigmatism | up to 6 months
  The safety index (unitless parameter) is calculated as postoperative CDVA/ preoperative CDVA (both in decimal units).
The efficacy index of using 7 and 6.5 mm lenticule diameters SMILE to treat myopic astigmatism | up to 6 months
  The efficacy index (unitless parameter) is calculated as postoperative UDVA/ preoperative CDVA (both in decimal units).

SECONDARY OUTCOMES:
Refractive outcomes of using 7 and 6.5 mm lenticule diameters SMILE to treat myopic astigmatism. | up to 6 months
  To compare subjective refractive outcomes including spherical equivalent and residual astigmatism (in diopters) of SMILE procedure using 7 and 6.5 mm lenticule diameters SMILE to treat myopic astigmatism.
Visual acuity outcomes of using 7 and 6.5 mm lenticule diameters SMILE to treat myopic astigmatism. | up to 6 months
  To compare postoperative UDVA and CDVA (in logMAR) of SMILE procedure using 7 and 6.5 mm lenticule diameters SMILE to treat myopic astigmatism.
Contrast sensitivity outcomes of using 7 and 6.5 mm lenticule diameters SMILE to treat myopic astigmatism. | up to 6 months
  To compare postoperative photopic and mesopic contrast sensitivity (in log unit) at 3, 6, 12, and 18 cycles per degree of SMILE procedure using 7 and 6.5 mm lenticule diameters SMILE to treat myopic astigmatism. This will be done using the CSV1000E device (Good-Lite, Elgin, IL, USA)
Corneal curvature changes after SMILE procedure using 7 and 6.5 mm lenticule diameters SMILE to treat myopic astigmatism. | up to 6 months
  To compare postoperative corneal curvature in flattest and steepest meridia (in keratometric diopters) after SMILE procedure using 7 and 6.5 mm lenticule diameters SMILE to treat myopic astigmatism. This will be done using the Pentacam high resolution (HR) (Oculus Optikgeräte, Wetzlar, Germany).
Corneal structural changes after SMILE procedure using 7 and 6.5 mm lenticule diameters SMILE to treat myopic astigmatism. | up to 6 months
  To compare postoperative and central corneal and epithelial thickness (in micrometers) and standard deviation of epithelial thickness in different locations (in micrometers) after SMILE procedure using 7 and 6.5 mm lenticule diameters SMILE to treat myopic astigmatism. This will be done using the anterior segment OCT (Cirrus HD-OCT, Carl Zeiss Meditec, Jena, Germany)

CONTACTS AND LOCATIONS:
Locations (1):
- Al Watany Eye Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sekundo W, Kunert KS, Blum M. Small incision corneal refractive surgery using the small incision lenticule extraction (SMILE) procedure for the correction of myopia and myopic astigmatism: results of a 6 month prospective study. Br J Ophthalmol. 2011 Mar;95(3):335-9. doi: 10.1136/bjo.2009.174284. Epub 2010 Jul 3. PMID 20601657
- [Background] Zhang J, Wang Y, Wu W, Xu L, Li X, Dou R. Vector analysis of low to moderate astigmatism with small incision lenticule extraction (SMILE): results of a 1-year follow-up. BMC Ophthalmol. 2015 Jan 24;15:8. doi: 10.1186/1471-2415-15-8. PMID 25618419
- [Background] Ivarsen A, Hjortdal J. Correction of myopic astigmatism with small incision lenticule extraction. J Refract Surg. 2014 Apr;30(4):240-7. doi: 10.3928/1081597X-20140320-02. PMID 24702575
- [Background] Ganesh S, Brar S, Pawar A. Results of Intraoperative Manual Cyclotorsion Compensation for Myopic Astigmatism in Patients Undergoing Small Incision Lenticule Extraction (SMILE). J Refract Surg. 2017 Aug 1;33(8):506-512. doi: 10.3928/1081597X-20170328-01. PMID 28787514
- [Background] Pedersen IB, Ivarsen A, Hjortdal J. Changes in Astigmatism, Densitometry, and Aberrations After SMILE for Low to High Myopic Astigmatism: A 12-Month Prospective Study. J Refract Surg. 2017 Jan 1;33(1):11-17. doi: 10.3928/1081597X-20161006-04. PMID 28068441